CLINICAL TRIAL: NCT06412887
Title: Effects of Adding Force Control to a VR Game on Brain Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Fong Chin Su, Chair Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 112-181
Record Dates: First submitted 2024-04-25; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Healthy Aging
Keywords: Virtual Reality; functional near infrared spectroscopy

STUDY DESIGN:
Intervention Model Description: Subjects play the virtual reality game using the wfc input system followed by the wofc input system
Masking Description: The subjects were informed regarding which input system was to be used
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with force control (wfc) (Active Comparator): Users play the game using the conventional virtual reality input system with force control
  Interventions: Device: Virtual reality headset
- without force control (wofc) (Experimental): Users play the game using the conventional virtual reality input system
  Interventions: Device: Virtual reality headset

INTERVENTIONS:
Device: Virtual reality headset — Meta-Quest 2 virtual reality headset was used in this study

SUMMARY:
One of the major contributor for the lower quality of living in the aged population, is the reduction in hand function. To mitigate this, several virtual-reality based hand rehabilitation/training systems have been developed.

However, most of these systems are solely controlled by hand gestures, and do not incorporate the force between the fingertips. Which is not the case for grabbing things in real life. With that in mind, the researchers assumed that a virtual-reality based hand rehabilitation/training system that incorporates force control into its input can be more beneficial in terms of recovering one's hand function.

To test out this claim, subjects were recruited and tasked to play a game using both input systems (wfc and wofc), while their brain activity while using both input system was simultaneously recorded using functional near infrared spectroscopy and compared

ELIGIBILITY:
Inclusion Criteria:

* With normal vision or wearing prescription glass that can fit inside the Meta Quest 2 VR headset.
* Able to understand English, Chinese, or Taiwanese language.

Exclusion Criteria:

* Experiencing motion sickness after prolonged usage of VR headsets
* Having chronic diseases or injuries that can prevent them from participating in the experiment such as: hand injuries, missing fingers, blindness, deafness, hearing impairments, etc.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Oxygenated hemoglobin (HbO) | 1 hour
  The Oxygenated hemoglobin (HbO) was measured while the participants play the game under both conditions
Game performance1 (Amount of grasp initiated) | 1 hour
  This unitless metric counts the number of times the subject initiates a grasp while playing the game, a higher amount of grasp initiated signifies worst performance
Game performance2 (Memory task accuracy) | 1 hour
  This percentage is calculated by dividing the amount of correct response by the total amount of response. A larger perrcentage represents better performance

SECONDARY OUTCOMES:
Manual dexterity | 5 minutes
  The manual dexterity of each participant was measured using the Purdue Pegboard Test at the beginning of the experiment
Maximum voluntary pinch force | 5 minutes
  The maximum voluntary pinch force of each particapant were measured using the Jamar pinch dynamometer at the beginning of the experiment
Recall | 5 minutes
  The ability to recall information of each particapant was measured using the forward digit span test at the beginning of the experiment

CONTACTS AND LOCATIONS:
Overall Officials: Fong-Chin Su, PhD, Principal Investigator — Chair Professor
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kivell TL. Evidence in hand: recent discoveries and the early evolution of human manual manipulation. Philos Trans R Soc Lond B Biol Sci. 2015 Nov 19;370(1682):20150105. doi: 10.1098/rstb.2015.0105. PMID 26483538
- [Background] Vergara M, Sancho-Bru JL, Gracia-Ibanez V, Perez-Gonzalez A. An introductory study of common grasps used by adults during performance of activities of daily living. J Hand Ther. 2014 Jul-Sep;27(3):225-33; quiz 234. doi: 10.1016/j.jht.2014.04.002. Epub 2014 Apr 21. PMID 24878351
- [Background] Smaby N, Johanson ME, Baker B, Kenney DE, Murray WM, Hentz VR. Identification of key pinch forces required to complete functional tasks. J Rehabil Res Dev. 2004 Mar;41(2):215-24. doi: 10.1682/jrrd.2004.02.0215. PMID 15558375
- [Background] Kurillo G, Gregoric M, Goljar N, Bajd T. Grip force tracking system for assessment and rehabilitation of hand function. Technol Health Care. 2005;13(3):137-49. PMID 15990417
- [Background] Magni NE, McNair PJ, Rice DA. Impairments in grip and pinch force accuracy and steadiness in people with osteoarthritis of the hand: A case-control comparison. Musculoskelet Sci Pract. 2021 Oct;55:102432. doi: 10.1016/j.msksp.2021.102432. Epub 2021 Jul 22. PMID 34333399
- [Background] Strote C, Golz C, Stroehlein JK, Haase FK, Koester D, Reinsberger C, Vieluf S. Effects of force level and task difficulty on force control performance in elderly people. Exp Brain Res. 2020 Oct;238(10):2179-2188. doi: 10.1007/s00221-020-05864-1. Epub 2020 Jul 13. PMID 32661649
- [Background] Howard, M. C. (2017). A meta-analysis and systematic literature review of virtual reality rehabilitation programs. Computers in Human Behavior, 70, 317-327. https://doi.org/10.1016/j.chb.2017.01.013
- [Background] Pereira, M. F., Prahm, C., Kolbenschlag, J., Oliveira, E., & Rodrigues, N. F. (2020). A Virtual Reality Serious Game for Hand Rehabilitation Therapy. 2020 IEEE 8th International Conference on Serious Games and Applications for Health (SeGAH), 1-7. https://doi.org/10.1109/SeGAH49190.2020.9201789
- [Background] Vanbellingen T, Filius SJ, Nyffeler T, van Wegen EEH. Usability of Videogame-Based Dexterity Training in the Early Rehabilitation Phase of Stroke Patients: A Pilot Study. Front Neurol. 2017 Dec 8;8:654. doi: 10.3389/fneur.2017.00654. eCollection 2017. PMID 29276499
- [Background] Friedman N, Chan V, Reinkensmeyer AN, Beroukhim A, Zambrano GJ, Bachman M, Reinkensmeyer DJ. Retraining and assessing hand movement after stroke using the MusicGlove: comparison with conventional hand therapy and isometric grip training. J Neuroeng Rehabil. 2014 Apr 30;11:76. doi: 10.1186/1743-0003-11-76. PMID 24885076
- [Background] Bae SJ, Jang SH, Seo JP, Chang PH. The Optimal Speed for Cortical Activation of Passive Wrist Movements Performed by a Rehabilitation Robot: A Functional NIRS Study. Front Hum Neurosci. 2017 Apr 20;11:194. doi: 10.3389/fnhum.2017.00194. eCollection 2017. PMID 28473763
- [Background] Zheng J, Ma Q, He W, Huang Y, Shi P, Li S, Yu H. Cognitive and motor cortex activation during robot-assisted multi-sensory interactive motor rehabilitation training: An fNIRS based pilot study. Front Hum Neurosci. 2023 Feb 9;17:1089276. doi: 10.3389/fnhum.2023.1089276. eCollection 2023. PMID 36845877
- [Background] Xia W, Dai R, Xu X, Huai B, Bai Z, Zhang J, Jin M, Niu W. Cortical mapping of active and passive upper limb training in stroke patients and healthy people: A functional near-infrared spectroscopy study. Brain Res. 2022 Aug 1;1788:147935. doi: 10.1016/j.brainres.2022.147935. Epub 2022 Apr 29. PMID 35500604
- [Background] Hummel, J., Dodiya, J., Wolff, R., Gerndt, A., & Kuhlen, T. (2013). An evaluation of two simple methods for representing heaviness in immersive virtual environments. 2013 IEEE Symposium on 3D User Interfaces (3DUI), 87-94. https://doi.org/10.1109/3DUI.2013.6550202